CLINICAL TRIAL: NCT00878163
Title: Phase I Trial of the Combination of Vismodegib GDC-0449 and Erlotinib +/- Gemcitabine
Brief Title: GDC-0449 and Erlotinib Hydrochloride With or Without Gemcitabine Hydrochloride in Treating Patients With Metastatic Pancreatic Cancer or Solid Tumors That Cannot Be Removed by Surgery
Status: Active, not recruiting | Phase: Phase 1 | Type: Interventional
Sponsor: National Cancer Institute (NCI) (NIH)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: NCI-2011-01400; NCI-2011-01400 (Registry Identifier: CTRP (Clinical Trial Reporting Program)); CDR0000638302; MAYO-MC0811; MC0811 (Other: Mayo Clinic in Rochester); 8231 (Other: CTEP); P30CA015083 (NIH); P50CA102701 (NIH); U01CA069912 (NIH)
Record Dates: First submitted 2009-04-07; First posted 2009-04-08 (Estimated); Last update posted 2025-09-09 (Actual); Status verified 2025-09

CONDITIONS: Adult Solid Neoplasm; Pancreatic Acinar Cell Carcinoma; Pancreatic Ductal Adenocarcinoma; Recurrent Pancreatic Carcinoma; Stage IV Pancreatic Cancer AJCC v6 and v7
MeSH Terms: conditions — Pancreatic Neoplasms | interventions — Erlotinib Hydrochloride; Gemcitabine; HhAntag691

ARMS (1):
- Treatment (vismodegib, erlotinib hydrochloride, gemcitabine) (Experimental): Patients receive Hedgehog antagonist GDC-0449 PO QD and erlotinib hydrochloride PO QD on days 1-28. Some patients also receive gemcitabine hydrochloride IV over 30 minutes on days 1, 8, and 15. Courses repeat every 28 days in the absence of disease progression or unacceptable toxicity.
  Interventions: Other: Diagnostic Laboratory Biomarker Analysis; Drug: Erlotinib Hydrochloride; Drug: Gemcitabine Hydrochloride; Drug: Vismodegib

INTERVENTIONS:
Other: Diagnostic Laboratory Biomarker Analysis — Correlative studies
Drug: Erlotinib Hydrochloride — Given PO
  Other Names: CP 358; CP-358; Cp-358,774; CP358; OSI 774; OSI-774; OSI774; Tarceva
Drug: Gemcitabine Hydrochloride — Given IV
  Other Names: dFdCyd; Difluorodeoxycytidine Hydrochloride; Gemcitabine HCI; Gemzar; LY 188011; LY-188011; LY188011
Drug: Vismodegib — Given PO
  Other Names: Erivedge; GDC 0449; GDC-0449; GDC0449; Hedgehog Antagonist GDC-0449

SUMMARY:
This phase I trial is studying the side effects and best dose of erlotinib hydrochloride when given together with GDC-0449 with or without gemcitabine hydrochloride in treating patients with metastatic pancreatic cancer or solid tumors that cannot be removed by surgery. Drugs used in chemotherapy, such as GDC-0449 and gemcitabine hydrochloride, work in different ways to stop the growth of tumor cells, either by killing the cells or by stopping them from dividing. Erlotinib hydrochloride may stop the growth of tumor cells by blocking some of the enzymes needed for cell growth. Giving GDC-0449 together with erlotinib hydrochloride with or without gemcitabine hydrochloride may kill more tumor cells.

DETAILED DESCRIPTION:
PRIMARY OBJECTIVES:

I. To determine the maximum tolerated dose of erlotinib hydrochloride and Hedgehog antagonist GDC-0449 with or without gemcitabine hydrochloride in patients with unresectable solid tumors.

SECONDARY OBJECTIVES:

I. To describe the adverse events profile associated with these treatment regimens.

II. To describe the responses in patients treated with these regimens. III. To assess the effect of erlotinib hydrochloride and Hedgehog antagonist GDC-0449 on selected biomarkers in circulating tumor cells and tumor biopsy samples from patients with metastatic pancreatic cancer.

IV. To assess the effect of erlotinib hydrochloride and Hedgehog antagonist GDC-0449 on fludeoxyglucose F 18 positron emission tomography imaging in patients with metastatic pancreatic cancer.

V. To study the association between clinical (toxicity and/or tumor response or activity) and biologic (pharmacodynamic) results associated with erlotinib hydrochloride and Hedgehog antagonist GDC-0449 in patients with metastatic pancreatic cancer.

OUTLINE: This is a dose-escalation study of erlotinib hydrochloride.

Patients receive Hedgehog antagonist GDC-0449 orally (PO) once daily (QD) and erlotinib hydrochloride PO QD on days 1-28. Some patients also receive gemcitabine hydrochloride IV over 30 minutes on days 1, 8, and 15. Courses repeat every 28 days in the absence of disease progression or unacceptable toxicity.

Patients treated at the maximum tolerated dose undergo fludeoxyglucose F 18 positron emission tomography at baseline and on day 28. These patients also undergo tumor tissue and blood sample collection at baseline and periodically during study for correlative laboratory studies. Samples are analyzed for tyrosine phosphorylated or total MAP-K, EGFR, AKT, and other potential biomarkers of activity/response and for levels of genes transcriptionally activated (e.g., BCL-2, GLI, BFL-1/A1, 4-1BB, PTC1) by immunofluorescence, IHC, and quantitative-PCR.

After completion of study therapy, patients are followed at 3 months.

ELIGIBILITY:
Inclusion Criteria:

* Histologic proof of a solid tumor that is now unresectable, not amenable to any other standard therapies, or patient refuses standard therapy

  * Metastatic adenocarcinoma of the pancreas amenable to biopsies (cohort II MTD only)
* Absolute neutrophil count (ANC) >= 1,500/μL
* Platelets >= 100,000/μL
* Total bilirubin =< upper limit of normal (ULN)
* Aspartate aminotransferase (AST) =< 3 times upper limit of normal (ULN)
* Creatinine =< 1.5 times ULN
* Hemoglobin >= 9.0 g/dL
* International Normalized Ratio (INR) within normal limits (for patients treated at the MTD)
* Ability to provide informed consent
* Willingness to return to Mayo Clinic for follow up
* Life expectancy >= 12 weeks
* Willingness to provide the biologic specimens as required by the protocol
* Negative serum pregnancy test done =< 7 days prior to registration
* Eastern Cooperative Oncology Group (ECOG) performance status (PS) 0-2
* Able to swallow or have medication administered through a G-tube and absorb the medication
* Participant agrees to use an acceptable form of contraception; acceptable forms of contraception:

  * Latex condom (always used with spermicide)
  * Diaphragm (always used with spermicide)
  * Cervical cap (always used with spermicide)

Acceptable forms of secondary contraceptions, when used along with a barrier method:

* Hormonal contraception methods, including pills, patches, rings, or injections except progestin-only containing pills (i.e. "Mini-pill")
* Tubal ligation
* Partner's vasectomy
* Intrauterine device (IUD) (non-progesterone T)
* Vaginal sponge (containing spermicide)
* 100% commitment to abstinence

Unacceptable forms of contraception for women of childbearing potential:

* Oral contraception containing progestins only
* IUD progesterone T
* Female condom
* Natural family planning (rhythm method) or breastfeeding
* Fertility awareness
* Withdrawal
* Cervical shield

  * Willing to abstain from smoking
  * Willing to complete a daily pill diary

Exclusion Criteria:

* Known standard therapy for the patient's disease that is potentially curative or definitely capable of extending life expectancy
* Uncontrolled intercurrent illness including, but not limited to, ongoing or active infection, symptomatic congestive heart failure, unstable angina pectoris, cardiac arrhythmia, or psychiatric illness/social situations that would limit compliance with study requirements
* Any of the following prior therapies:

  * Chemotherapy =< 4 weeks prior to registration
  * Mitomycin C/nitrosoureas =< 6 weeks prior to registration
  * Immunotherapy =< 4 weeks prior to registration
  * Biologic therapy =< 4 weeks prior to registration
  * Radiation therapy =< 4 weeks prior to registration
  * Radiation to > 25% of bone marrow
* Failure to fully recover from acute, reversible effects of prior therapy regardless of interval since last treatment
* New York Heart Association classification III or IV
* Seizure disorder
* Central nervous system (CNS) metastases if not stable for at least 2-3 months based on imaging, clinical assessment, and use of steroids, or seizure disorder
* Pregnant women
* Nursing women
* Men or women of childbearing potential who are unwilling to employ adequate contraception until 12 months after last study drug dose
* Other concurrent chemotherapy, immunotherapy, radiotherapy, or any ancillary therapy considered investigational (utilized for a non-Food and Drug Administration [FDA]-approved indication and in the context of a research investigation)
* Current therapy with a CYP3A4 inhibitor or inducer
* Immunocompromised patients (other than that related to the use of corticosteroids) including patients receiving highly active antiretroviral therapy (HAART) treatment
* Receiving any other investigational agent which would be considered as a treatment for the primary neoplasm
* Active other malignancy, excepting non-melanotic skin cancer or carcinoma-in-situ of the cervix; if there is a history of prior malignancy, they must not be receiving other specific treatment (other than hormonal therapy) for their cancer
* History of myocardial infarction =< 6 months, or congestive heart failure requiring use of ongoing maintenance therapy for life-threatening ventricular arrhythmias
* Abnormalities of the cornea based on history (e.g., dry eye syndrome, Sjogren's syndrome), congenital abnormality (e.g., Fuch's dystrophy), abnormal slit-lamp examination using a vital dye (e.g., fluorescein, Bengal Rose), and/or an abnormal corneal sensitivity test (Schirmer test or similar tear production test)
* More than 2 prior chemotherapy regimens for the current metastatic malignancy; full dose chemotherapy used in conjunction with concurrent radiation therapy will be included as prior therapy; Note: prior hormonal therapy (e.g. leuprolide, aromatase inhibitors, tamoxifen) will be allowed and not included as a prior chemotherapy
* Previous therapy with a hedgehog inhibitor

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 55 (Actual)
Dates: Start 2009-03-31 (Actual); Primary Completion 2013-01-22 (Actual); Study Completion 2026-03-06 (Estimated)

PRIMARY OUTCOMES:
Maximum tolerated dose of erlotinib hydrochloride defined as the dose level below the lowest dose that induces dose-limiting toxicity in at least one-third of patients | 28 days
  DLT will be defined as an adverse event, according to CTCAE version 3.0, attributed (definitely, probably, or possibly to the study treatment.

SECONDARY OUTCOMES:
Adverse events as assessed by NCI CTCAE v3.0 | Up to 3 months after completion of study treatment
  The number and severity of all adverse events (overall, and by dose-level) will be tabulated and summarized.
Toxicity, defined as adverse events that are classified as either possibly, probably, or definitely related to study treatment, graded using the NCI CTCAE version 3.0 | Up to 3 months after completion of study treatment
Response as assessed by modified RECIST criteria | Up to 3 months after completion of study treatment
  Summarized by simple descriptive summary statistics delineating complete and partial responses as well as stable and progressive disease.
Time until treatment related grade 3+ toxicity | Up to 3 months after completion of study treatment
Time until hematologic nadirs (WBC, ANC, platelets) | Up to 3 months after completion of study treatment
Time to progression | Up to 3 months after completion of study treatment
Time to treatment failure | From registration to documentation of progression, unacceptable toxicity, or refusal to continue participation by the patient, assessed up to 3 months after completion of study treatment

CONTACTS AND LOCATIONS:
Overall Officials: Charles Erlichman, Principal Investigator — Mayo Clinic
Locations (4):
- United States (4):
  - Mayo Clinic in Arizona, Scottsdale, Arizona
  - Mayo Clinic in Florida, Jacksonville, Florida
  - Orlando Health Cancer Institute, Orlando, Florida
  - Mayo Clinic in Rochester, Rochester, Minnesota